CLINICAL TRIAL: NCT04256616
Title: Immunogenic Cell Death as a Novel Mechanism of Mitomycin C Activity in Bladder Cancer
Acronym: ICH-MIM-01
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Istituto Clinico Humanitas (Other)
Responsible Party: Principal Investigator, Michele Tedeschi, Head of Clinical Research, Istituto Clinico Humanitas
Other Study IDs: 2041
Record Dates: First submitted 2020-02-03; First posted 2020-02-05 (Actual); Last update posted 2020-07-07 (Actual); Status verified 2020-07

CONDITIONS: Bladder Cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Bladder cancer patients: 80 patients with carcinoma of the bladder; divided in 20 patients Ta (low grade), 20 patients Ta/T1 (high grade) and 20 patients T2. Only for liquid samples collection we will include 20 CIS (carcinoma in situ) patients
  Interventions: Other: This is an observational study that does not concern a direct intervention on patients and control subjects and does not interfere with the clinical management of patients.
- Controls- Healthy subjects: 30 age and sex-matched subjects not suffering from carcinoma of the bladder, already hospitalized in ICH; we expect to enroll 24 males and 6 females of which 10 of 40- 60 years old, 10 of 60-70 years old, 10 of >70 years old.
  Interventions: Other: This is an observational study that does not concern a direct intervention on patients and control subjects and does not interfere with the clinical management of patients.

INTERVENTIONS:
Other: This is an observational study that does not concern a direct intervention on patients and control subjects and does not interfere with the clinical management of patients. — urine collection: DNA is isolated from urine samples (catheterized, washout, midstream) and the 16S rRNA gene is sequenced.
  Specimen collection: Specimens collected during TURBT are selected by a pathologist and trasferred to the laboratory. The tissues are treated ex vivo with MMC.

SUMMARY:
The principal objective of this study consists in the assessment of Immunogenic Cell Death (ICD) induction in neoplastic tissues derived from bladder cancer patients treated ex vivo with Mitomycin C (MMC). The evaluation is performed using cellular and molecular analyses of treated versus untreated samples derived from the same patient

DETAILED DESCRIPTION:
Urothelial or transitional cell carcinoma of the bladder is the fourth most common cancer in males worldwide, with about 60-80% of newly diagnosed patients having non-muscle-invasive bladder cancer (NMIBC). NMIBC management consist in transurethral resection of bladder tumor (TURBT) followed by adjuvant intravesical treatment with the chemotherapeutic agent Mitomycin C (MMC) or the immunotherapy bacillus Calmette-Guérin. These therapies result in low progression rates, but are not efficacious in all patients, leading to high tumor recurrence. Immunogenic cell death (ICD) may be one of the mechanisms of action of MMC intravesical therapy in bladder cancer.

The primary objective of the study is to evaluate whether MMC is able to trigger ICD in patient-derived neoplastic tissues. As secondary targets we aim to:

1. identify an expression profile that is common to all tumors that undergo ICD upon MMC treatment ('ICD signature'),
2. asses the genetic and environmental factors- urinary microbiome composition- responsible for MMC treatment efficacy,
3. evaluate whether ICD induction correlates with clinical staging and response (clinical endpoints for MMC-treated patients are recurrence at three month and one year after enrollment).

ELIGIBILITY:
Inclusion Criteria:

- Male and females, > 40 years old

For bladder cancer patients:

- bladder cancer patients- patinets with first tumor occurrence or patient with a recurrence after more than 2 years from the removal of the prior malignancy

Exclusion Criteria:

* Treated with immunomodulatory agents at time of enrollment or in the two months before enrollment
* Treated with antibiotics at time of enrollment or during the month before enrollment
* Positive history of sexually transmitted diseases
* Urinary infection ongoing or recent (during the three months before enrollment)
* Suffering from chronic intestinal inflammation

ONLY for controls:

* Treated with immunomodulatory agents at time of enrollment or in the two months before enrollment
* Treated with antibiotics at time of enrollment or during the month before enrollment
* Positive history of sexually transmitted diseases
* Urinary infection ongoing or recent (during the three months before enrollment)
* Suffering from chronic intestinal inflammation

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 80 patients with carcinoma of the bladder; divided in 20 patients Ta (low grade), 20 patients Ta/T1 (high grade) and 20 patients T2. Only for liquid samples collection we will include 20 CIS (carcinoma in situ) patients.
  30 age and sex-matched subjects not suffering from carcinoma of the bladder, already hospitalized in ICH; we expect to enroll 24 males and 6 females of which 10 of 40- 60 years old, 10 of 60-70 years old, 10 of >70 years old.
Sampling Method: Non-Probability Sample
Enrollment: 110 (Estimated)
Dates: Start 2018-06-27 (Actual); Primary Completion 2020-09-01 (Estimated); Study Completion 2020-09-30 (Estimated)

PRIMARY OUTCOMES:
MMC-induced ICD | 3 years
  The main aim of this study is to evaluate whether MMC is able to trigger ICD in patient-derived neoplastic tissues.

SECONDARY OUTCOMES:
ICD signature analyzed by RNAseq analysis | 3 years
  Identify an expression profile that is common to all tumors that undergo ICD upon MMC treatment ('ICD signature')
Microbiota study | 3 years
  Verify the existance of urinary microbiome using catheterized urines and identify changes in urinary microbiome composition correlating with bldder cancer, MMC efficacy and staging/progression of the disease

CONTACTS AND LOCATIONS:
Locations (1):
- Humanitas reseach hospital (ICH), Rozzano, Milan, Italy

IPD SHARING:
Plan to Share IPD: No
Research outcome

REFERENCES:
- [Derived] Oresta B, Pozzi C, Braga D, Hurle R, Lazzeri M, Colombo P, Frego N, Erreni M, Faccani C, Elefante G, Barcella M, Guazzoni G, Rescigno M. Mitochondrial metabolic reprogramming controls the induction of immunogenic cell death and efficacy of chemotherapy in bladder cancer. Sci Transl Med. 2021 Jan 6;13(575):eaba6110. doi: 10.1126/scitranslmed.aba6110. PMID 33408185